CLINICAL TRIAL: NCT06462118
Title: A Phase 1, Open-Label, Randomized, Single Dose Study to Evaluate the Effect of Injection Site on the Pharmacokinetics of Astegolimab in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of Injection Site on PK of Astegolimab in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GP45400
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — astegolimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment A (Experimental): Participants will receive one subcutaneous (SC) dose in the abdomen.
  Interventions: Drug: Astegolimab
- Treatment B (Experimental): Participants will receive one subcutaneous (SC) dose in the thigh.
  Interventions: Drug: Astegolimab
- Treatment C (Experimental): Participants will receive one subcutaneous (SC) dose in the upper arm.
  Interventions: Drug: Astegolimab

INTERVENTIONS:
Drug: Astegolimab — Participants will receive one SC dose of astegolimab in the abdomen, upper arm, or thigh.

SUMMARY:
The main objective is to study how astegolimab may behave in the body when injected subcutaneously into the abdomen, thigh, or upper arm in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Body weight of ≥50 kg to ≤110 kg with body mass index (BMI) range 18.0 to 30.0 kg/m2 (inclusive) at screening

Exclusion Criteria:

* History of significant hypersensitivity or severe allergic reaction, including anaphylaxis, to any drug compound, food, or other substance
* Any immunization or vaccination 14 days prior to the Check-in (Day -1) or plans to obtain any immunization or vaccination within 30 days after the Check-in
* Any surgical procedure (except for minor surgeries) within 28 days prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
* Donation of blood from 30 days prior to screening through study completion or end of trial, inclusive, or of plasma from 2 weeks prior to screening through study completion or end of trial, inclusive
* History of immunodeficiency, including but not limited to, human immunodeficiency virus (HIV) infection
* History of active or untreated latent tuberculosis
* History of malignancy within 5 years prior to screening, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or Stage I uterine cancer
* Unstable cardiac disease, myocardial infarction, or New York Heart Association Class 3 or 4 heart failure within 12 months prior to screening
* History or presence of clinically significant ECG abnormalities at screening or check-in (Day -1)
* Positive for Hepatitis B or Hepatitis C (HCV)
* Tattoo(s) or scarring at or near the site of injection (abdomen, front and middle thigh, or upper arm) or any other condition which may interfere with the injection site examination (as determined by the Investigator)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2024-06-17 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-22 (Actual)

PRIMARY OUTCOMES:
Area under the curve from Hour 0 to the time of last measurable concentration (AUC0-t) of astegolimab | Approximately 85 days
AUC extrapolated to infinity (AUC0-infinity) of astegolimab | Approximately 85 days
Maximum serum concentration (Cmax) of astegolimab | Approximately 85 days

SECONDARY OUTCOMES:
Relative bioavailability (F%) for thigh injection of astegolimab | Approximately 85 days
F% for upper arm injection of astegolimab | Approximately 85 days
Half-life (T1/2) of astegolimab | Approximately 85 days
Apparent systemic clearance (CL/F) of astegolimab | Approximately 85 days
Apparent volume of distribution during the terminal elimination phase (Vz/F) of astegolimab | Approximately 85 days
Time to maximum serum concentration (Tmax) of astegolimab | Approximately 85 days
Incidence of anti-drug antibodies (ADAs) | Approximately 85 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- United States (3):
  - Covance Research Unit - Daytona, Daytona Beach, Florida
  - Covance Research Unit - Dallas, Dallas, Texas
  - Covance Clinical Research Unit, Inc, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No